CLINICAL TRIAL: NCT04742881
Title: Low Impact Laparoscopic in Colorectal Resection: a Randomized Trial Comparing Low Pneumoperitoneum Pressure Plus Microsurgery Versus Low Pneumoperitoneum Alone
Brief Title: Low Impact Laparoscopic in Colorectal Resection - PAROS2
Acronym: PAROS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2020/30
Record Dates: First submitted 2021-01-22; First posted 2021-02-08 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Malignant or Benign Pathology
Keywords: Colorectal pathology; Laparoscopic; Microsurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low pressure + microsurgical instruments (Experimental): Low pressure pneumoperitoneum ((≤ 8 mmHg) and use of microsurgical instruments (3mm and 5mm instruments)
  Interventions: Procedure: Low pressure + microsurgical instruments
- Low pressure + standard instruments (Active Comparator): Low pressure pneumoperitoneum ((≤ 8 mmHg) and use of standard instruments (5mm and 10mm instruments)
  Interventions: Procedure: Low pressure + standard instruments

INTERVENTIONS:
Procedure: Low pressure + microsurgical instruments — Low pressure pneumoperitoneum ((≤ 8 mmHg) and use of microsurgical instruments (3mm and 5mm instruments)
  Arms: Low pressure + microsurgical instruments
Procedure: Low pressure + standard instruments — Low pressure pneumoperitoneum ((≤ 8 mmHg) and use of standard instruments (5mm and 10mm instruments)
  Arms: Low pressure + standard instruments

SUMMARY:
To improve post-operative recovery, the concept of Low Impact Laparoscopy was developed in colo-rectal surgery with associating low-pressure pneumoperitoneum and microlaparoscopic surgery. A phase III double-blind, prospective, randomized, controlled, multi-centric trial is designed in the aim to assess the impact of low-pressure pneumoperitoneum with microlaparoscopic instruments on post-operative pain at 24 hours without taking opioids. It is compared with low-pressure laparoscopy with classical laparoscopic instruments in patients undergoing colorectal surgeries.

DETAILED DESCRIPTION:
Laparoscopy is the gold standard in colorectal surgery with many benefits in term of morbidity, post-operative pain and analgesic consumption. However the pneumoperitoneum created for the laparoscopy has several negatives impact and limits (specific pain following abdominal distension, visibility, physiological repercussion).

To improve recovery after colorectal laparoscopic surgery it was realized a first study (PAROS) which showed that low-pressure laparoscopic colectomy for benign or malign disease was feasible and safe with shorter length of stay and decrease post-operative pain with reduction of analgesic consumption.

Minimally invasive technics like microlaparoscopic surgery, developed last years had also an impact by decreasing post operative pain. The Low Impact Laparoscopy concept was developed in colo-rectal surgery with the association of low-pressure pneumoperitoneum and microlaparoscopic surgery.

The aim of the study is to assess the impact of low-pressure pneumoperitoneum with microlaparoscopic instruments on post-operative pain without taking opioids, compared with low-pressure laparoscopy with classical laparoscopic instruments in patients undergoing colorectal surgeries.

The design of this study is a phase III double-blind, prospective, randomized, controlled, multi-centric trial. The primary endpoint is the rate of patients with postoperative pain defined 24h after the end of the intervention by visual analog scale (VAS) ≤ 3 without taking opioids (analgesics level II or III). Secondary outcomes are operating time, conversion rate in normal pressure laparoscopy or in laparotomy, morbidity at 3 months, quality of oncological surgery, length of stay, impact of microlaparoscopic instruments of aesthetic appearance at 3 months.

The primary end point will be assessed at 24h after the end of the surgery by a blind nurse evaluating the pain intensity. After discharge of the hospital, patients will be followed with postoperative consultation at 1 month and 3 month.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled colectomy for malignant or benign pathology
* Right colon: ileocecal resection, right colectomy, right colectomy extended to the middle of the transverse
* Left colon: sigmoidectomy, left colectomy
* Rectal resection without stoma for cancer of the upper rectum
* Patient operable by laparoscopy (classic or robot assisted for the Standard group)
* Age ≥ 18 years old
* Patient affiliated to a social security system or beneficiary of the same
* Informing the patient and obtaining free, informed and written consent, signed by the patient and his investigator

Exclusion Criteria:

* Laparotomy procedure
* Patients with electronic implant (ex : pacemaker)
* Total or Subtotal Colectomy
* Transverse segmental colectomy
* Left angular colectomy
* Proctectomy with stoma or Total Coloproctectomy
* Patient with stoma
* Probable realization of a stoma during the operation
* Procedure associated with colorectal surgery (except appendectomy or liver biopsy)
* Crohn's disease, Hemorrhagic Rectocolitis (UC)
* Sigmoiditis
* EVA before surgery> 3
* BMI ≥ 30
* ASA > 3
* History of laparotomy
* Emergency surgery
* Pelvic Sepsis or Preoperative Fistula
* Pregnant woman, likely to be, or breastfeeding
* Persons deprived of their liberty or under measure of judicial protection (curatorship or guardianship) or unable to give their consent
* Inability to undergo medical monitoring of the trial for geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with pain at 24 hours after the end of the intervention by NRS ≤ 3 without taking opioids (without pain reliever 2 and 3) | At 24 hours after the end of surgery
  Pain is evaluated with the Numeric Rating Scale (NRS, from 0 (no pain) to 10 (hurts worst)

SECONDARY OUTCOMES:
Operating time | During surgery
Conversion rate in normal pressure laparoscopy and or in laparotomy | During surgery
Intraoperative analgesia nociception index (ANI) | During surgery
Peri-operative cardiovascular and respiratory components | During surgery
Time to resume transit and gas | An average of 5 days after the surgery
Number of patients with medical and/or surgical morbidity | From the end of surgery until 3 months of follow-up
  To analyse the cumulative morbidity at 30 days after surgery and at 3 months of follow-up according to the Clavien-DINDO classification
Number of patients with R0 resection | During surgery
  Rate of curative surgery R0 resection for oncologic surgery
Number of lymph nodes examined | During surgery
  Number of lymph nodes examined by the pathologist for oncologic surgery
Length of stay in hospital | From surgery to the end of the hospitalization (max 30 days)
Number of patients with pain at 30 days | From the end of the surgery until 30 days of follow up
  Pain was evaluated with the Numeric Rating Scale during hospital stay and until 30 days using a patient subject diary every day and immediately before each use of pain medication
Number of patients taking analgesics until 30 days | From the end of the surgery until 30 days of follow up
  To analyse the rate of analgesics using a patient subject diary
Impact of microsurgical instruments on the aesthetic appearance | 30 days after surgery and 3 months of follow up
  Rate of scar satisfaction at 30days and at 3 months after surgery
Mean score of the EQ-5D-5L Quality of life | From randomization until 3 months of follow up
  Health related quality of life will be assessed using the Short Form EQ-5D-5L Health Survey questionnaire. The EQ-5D-5L is a generic health status measurement instrument. It is made up of 5 questions and a visual scale. A question for each of the following aspects: mobility, the ability to wash and dress, daily activities, discomfort and pain, anxiety as well as a score for the patient's perception of the quality of life. The questionnaire is administered the day before the surgery and 1 month and 3 months after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LAURENT, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- France (3):
  - CH de la Côte Basque, Bayonne
  - CHU Bordeaux, Bordeaux
  - Ch Libourne, Libourne

REFERENCES:
- [Derived] Marichez A, Eude A, Martenot M, Celerier B, Capdepont M, Rullier E, Denost Q, Fernandez B. Low-impact laparoscopy in colorectal resection-A multicentric randomised trial comparing low-pressure pneumoperitoneum plus microsurgery versus low-pressure pneumoperitoneum alone: The PAROS II trial. Colorectal Dis. 2023 Dec;25(12):2403-2413. doi: 10.1111/codi.16787. Epub 2023 Oct 27. PMID 37897108